CLINICAL TRIAL: NCT04287062
Title: Examining the Role of the Orexin System in Sleep and Stress in Persons With Opioid Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00223942; U01HL150835 (NIH)
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Sleep Disturbance; Opioid-use Disorder
MeSH Terms: conditions — Parasomnias; Opioid-Related Disorders | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo sleep medication (2 placebo oral capsules)
  Interventions: Drug: Placebos
- Suvorexant (Active Comparator): Sleep medication (20mg suvorexant; 2 10mg capsules; patients can self-titrate to 1 10mg capsule)
  Interventions: Drug: Suvorexant

INTERVENTIONS:
Drug: Suvorexant — Dual orexin receptor antagonist
  Arms: Suvorexant
Drug: Placebos — Weight and color matched placebo
  Arms: Placebo

SUMMARY:
This study is designed to elucidate the role of the orexin neurotransmitter system in sleep disturbance and circadian rhythms of stress that might in turn influence relapse behaviors in persons on medication-assisted treatments (MAT) who are in early recovery from opioid use disorder (OUD). Briefly, the study will enroll recently abstinent OUD patients (N=200) maintained on either extended-release naltrexone (XR-NTX), buprenorphine, or methadone. Within each MAT group, participants will be randomized to either suvorexant or placebo. The study is expected to have a 20% treatment attrition rate which will result in N=160 completers in the entire study. Patients will be recruited from and treated at Ashley Addiction Treatment, Addiction Treatment Services at Johns Hopkins Bayview Medical Center, Man Alive, or community providers.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 21-65, inclusive.
* Past 30-day sleep disturbance as evidenced by a Pittsburgh Sleep Quality Index Total Score >5.
* Enrolled in either outpatient methadone-maintenance, buprenorphine-maintenance, or XR-NTX treatment for OUD.
* Willingness to be maintained on a protocolized dose starting between 60-130mg methadone or 380mg XR-NTX for the duration of the study.
* At least two weeks of continuous abstinence from illicit opioids as evidenced by self-report and urine drug screens collected as part of routine care.
* Willing to comply with the study protocol, which will include weekly study visits, daily actigraphy and ecological momentary assessments.
* Use of birth control throughout study.
* Have no clinically significant chronic medical disorders or conditions that are judged by the investigators to prevent participation.

Exclusion Criteria:

* Serious mental illnesses that are unstable and could affect study participation (thought disorders, hallucinations, delusions, thoughts of harm to self/others).
* Current moderate to severe substance use disorder other than OUD.
* Current illicit stimulant use, including cocaine and methamphetamine.
* Pregnant or breast feeding.
* Have a known allergy to the study medications.
* Past 30-day prescribed use of suvorexant.
* Current use of a benzodiazepine or other schedule IV medication for insomnia.
* Use of Cytochrome P450 3A inhibitors.
* Current narcolepsy, sleep paralysis, or restless leg syndrome as assessed by medical history
* Apnea-hypopnea index > 30.
* Use of glucocorticoid medications and any medication that would alter the hypothalamic-pituitary-adrenal axis.
* Past 30-day suicidal behavior as assessed by the Columbia Suicide Severity Rating Scale (C-SSRS).
* Have circumstances that would interfere with study participation (e.g., impending jail; severe clinical issues).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-reported male or female
Enrollment: 138 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Total Sleep Time | 21 nights
  Mean total number of minutes slept per night as measured by actigraphy and self-reported sleep diary. Mean total sleep time will be collected over a seven-night period in weeks 1, 4, and 8 of the trial.
Total Wake Time After Sleep Onset | 21 nights
  Mean total number of minutes awake between initial sleep onset and final morning awakening, measured by actigraphy and self-reported sleep diary. Mean wake after sleep onset will be collected over a seven-night period in weeks 1, 4, and 8 of the trial.
Change in Perceived Stress Scale 4 (PSS-4) score | 21 days (collected over a seven-day period in weeks 1, 4, and 8 of the trial)
  Mean daily scores on the PSS-4 (a four item scale self-reported scale than measures stress using a 0-4 Likert scale; total range of PSS-4 scores is 0-16; lower scores indicate lower daily stress relative to higher scores, which indicate higher daily stress). Mean PSS-4 scores will be collected over a seven-day period in weeks 1, 4, and 8 of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Huhn, PhD, Principal Investigator — Johns Hopkins University
Locations (5):
- United States (5):
  - Man Alive Inc., Lane Treatment Center, Baltimore, Maryland
  - Addiction Treatment Services at Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Behavioral Pharmacology Research Unit at the Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Ashley Addiction Treatment, Bel Air, Maryland
  - Ashley Addiction Treatment, Elkton, Maryland

IPD SHARING:
Plan to Share IPD: No